CLINICAL TRIAL: NCT03378128
Title: Minimally Invasive Interval Debulking Surgery in Ovarian Cancer
Brief Title: Debulking Surgery in Ovarian Cancer
Acronym: MIID-SOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE9817
Record Dates: First submitted 2017-12-15; First posted 2017-12-19 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Malignant Neoplasm of Ovary; Malignant Neoplasm of Fallopian Tube; Malignant Neoplasm of Peritoneum
Keywords: debulking surgery; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diagnostic laparoscopic assessment after neoadjuvant chemo (Experimental): All patients will undergo a diagnostic laparoscopic assessment of disease following neoadjuvant chemotherapy
  Interventions: Procedure: Diagnostic laparoscopy

INTERVENTIONS:
Procedure: Diagnostic laparoscopy — The patient will initially undergo a diagnostic laparoscopy by a minimally invasive approach and entry method. The decision of which approach and entry to perform will be dictated by the primary surgeon of record's preference and their assessment of pre-operative patient factors. Once the primary surgeon determines the areas of macroscopic disease, he/she will make an assessment as to the need to convert to a laparotomy or continue laparoscopically. At the completion of the procedure, it will be noted whether an optimal cytoreduction (≤ 1 cm residual disease) or a sub-optimal cytoreduction (>1 cm residual disease) was performed.

SUMMARY:
The purpose of this study is to see if patients undergoing a laparoscopic surgery for removal of ovarian, fallopian tube, or primary peritoneal cancer following neoadjuvant chemotherapy (neoadjuvant- chemotherapy given before surgery) is feasible, safe, and provides similar outcomes as compared to undergoing a large abdominal incision. Minimally invasive, or laparoscopic, surgery is a type of surgery where only small incisions are made on the abdomen and surgical instruments are placed through these incisions to perform the surgery. This type of surgery has been shown to improve outcomes in many types of surgery, including in gynecologic cancer surgery. Specifically, researchers know that patients who have minimally invasive surgery have less pain after surgery, can go home quicker from the hospital, healing time is more rapid, and potentially this can translate into returning to chemotherapy sooner. Specifically, in ovarian, fallopian tube, and primary peritoneal cancer, minimally invasive surgery has not been used as much because these cancers can have tumors all throughout the inside of the abdomen (i.e. wide tumor burden) and located in areas that are sometimes not easily reachable with laparoscopic instruments. However, the reason patients receive neoadjuvant chemotherapy is to shrink the tumor/s to make the surgery less extensive and the recovery easier. It is unknown if minimally invasive surgery can be used in this setting and by studying this, the study team will be able to determine if patient outcomes are improved by implementing (using) this surgical technique.

DETAILED DESCRIPTION:
The objective of this study is to implement, evaluate, and further investigate the role of minimally invasive surgery in patients undergoing interval debulking following neoadjuvant chemotherapy in patients with advanced ovarian cancer.

Primary Objective:

Prospectively evaluate the feasibility and safety of the minimally invasive interval debulking approach

Secondary Objective(s)

1. Identify the patient population for which the minimally invasive interval debulking approach will offer comparable, if not improved, outcomes as the laparotomic interval debulking technique
2. Validate previously identified preoperative imaging computed tomography (CT) criteria and CA-125 values to predict optimal cytoreduction in laparotomic primary cytoreductive surgery and apply it towards the prediction of optimal cytoreduction (≤ 1 cm residual disease) following minimally invasive interval debulking surgery
3. Validate the previously identified laparoscopic scoring system for primary cytoreductive surgery and apply it towards the prediction of optimal cytoreduction (≤ 1 cm residual disease) following minimally invasive interval debulking surgery
4. Monitor the number of hospital days in the first 30 days postoperatively (length of stay after interval debulking including any days of readmission)
5. Evaluate the oncologic safety as it relates to time to return to chemotherapy in patients who undergo laparoscopic minimally invasive interval debulking surgery
6. Evaluate the complications as assessed by incidence of a composite of major complications and a second composite of minor complications

Study Design This will be a prospective pilot study to address feasibility and safety to identify a patient population amenable to this surgical approach. This will allow for the future trial to include randomization

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed advanced epithelial ovarian, fallopian tube, or primary peritoneal (≥ International Federation of Gynecology and Obstetrics (FIGO) Stage IIIC)
* Subjects must have received neoadjuvant chemotherapy (any number of cycles) with complete or partial response as assessed by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST) or CA 125 response by Gynecologic Cancer Intergroup (GCIG) criteria
* Performance status Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Severe cardiopulmonary disease precluding the use of the minimally invasive technique as deemed by Internal Medicine Preoperative Assessment, Consultant and Treatment (IMPACT)
* Inability to tolerate prolonged Trendelenburg position as deemed by anesthesiology
* Severe hip disease precluding the use of dorsolithotomy position
* Prior pelvic or abdominal radiation
* Clinically large pelvic masses reaching above the umbilicus
* Absence of a documented PR or CR according to RECIST 1.1 or CA 125 response by GCIG criteria to neoadjuvant chemotherapy
* Presence of parenchymal liver metastases on imaging
* Absence of baseline imaging studies (CT abdomen/pelvis and Chest x-ray minimum) both prior to beginning chemotherapy and following chemotherapy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who undergo minimally-invasive interval debulking surgery (MI-IDS) among all patients enrolled in the study | 1 day
  Feasibility measure
Percentage of patients experiencing grade 3 or 4 post-operative complications | 30 days post-surgery
  Accordion Severity Grading system with grade 3-4 scores. Grade 3 and 4 are severe complications or death. Severe complications are those requiring endoscopic or interventional radiologic procedures or re-operation as well as complications resulting in failure of 1 or more organ system. If fewer than 14% of patients have grade 3 or 4 complications, the surgery will be deemed safe.

SECONDARY OUTCOMES:
Percentage of patients with optimal cytoreductive surgery (=< 1cm of disease seen at completion of surgery) | 1 day
  Rate of optimal resection after interval debulking surgery is expected to be between 73%-81%
Proportion of patients who have a laparoscopy at the outset and remain laparoscopic throughout their surgery | 1 day
  If greater than 13 of the 50 patients planned to be enrolled on the study complete the laparoscopic surgery, the study will be deemed feasible
Length of hospital stay | Up to 30 days after surgery
  Time from the end of surgery to when the patient is discharged
Time to return to chemotherapy | 30 days after surgery
  From the time of surgery to when the patient returns to chemotherapy treatments. Shorter times between surgery and chemotherapy are positive outcomes
Score of the Bristow preoperative predictive index parameters | 1 day
  23 point index where higher scores indicate poorer outcomes
Score of Suidan preoperative predictive index parameters | 1 day
  17 point index where higher scores indicate poorer outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Chad Michener, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Atrium/Charlotte-Mecklenburg Hospital Authority, Charlotte, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Costales AB, Crane EK, Chambers L, Yao M, Chau D, Naumann WR, Debernardo R, Ricci S, Rose PG, Michener CM. Laparoscopic predictability of minimally invasive interval debulking in advanced ovarian cancer: The MIID-SOC trial. Gynecol Oncol. 2024 Jun;185:143-147. doi: 10.1016/j.ygyno.2024.02.019. Epub 2024 Feb 27. PMID 38417209